CLINICAL TRIAL: NCT02340390
Title: A PROSPECTIVE MULTI CENTER RANDOMIZED CONTROLLED TRIAL TO EVALUATE G7 Acetabular System With CoC ARTICULATION COMPARED TO EXCEED ABT Acetabular System With CoC ARTICULATION IN TOTAL HIP ARTHROPLASTY
Brief Title: G7 Acetabular System vs. Exceed ABT Acetabular System in THA
Acronym: G7
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ORTHO.CR.GH42
Record Dates: First submitted 2015-01-08; First posted 2015-01-16 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Osteoarthritis Arthritis; Rheumatoid Arthritis
Keywords: G7 Acetabular System
MeSH Terms: conditions — Joint Diseases; Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hip implant1 (Experimental): The Biomet G7 Acetabular System is a modular acetabular system, offering two types of acetabular shells. The shells are available in either a solid shell design, with an apical plug, or a limited hole with an apical plug and optional screw holes. Components are available in numerous designs and sizes intended for both primary and/or revision applications.
  Interventions: Device: G7
- Hip implant2 (Experimental): The Exceed ABT Acetabular System has been designed for cementless fixation and consists of an acetabular shell and an acetabular insert. The acetabular insert/bearing includes a tapered outer geometry that matches the inner geometry of the acetabular shell and an inner hemispherical geometry to suit the varying modular head diameters. Inserts/bearings are inserted into the acetabular shell intra-operatively and are available in varying sizes to match the acetabular shell diameters. The insert/bearings are available in Biolox Delta ceramic (CeramTec AG).
  Interventions: Device: Exceed ABT

INTERVENTIONS:
Device: G7 — The Biomet G7™ Acetabular System has been designed to provide more options to surgeons for treatment of patients needing total hip arthroplasty, while concurrently simplifying the surgical process with well-designed, modular components and corresponding instruments. The G7™ Acetabular System includes three liner types; ArComXL highly-crosslinked or E-1 Vitamin E-infused polyethylnene and a Biolox Delta (Ceramtec, Plochingen, Germany) ceramic liner.
  Arms: Hip implant1
Device: Exceed ABT — The Exceed ABT Acetabular System has been designed for cementless fixation and consists of an acetabular shell and an acetabular insert. The acetabular insert/bearing includes a tapered outer geometry that matches the inner geometry of the acetabular shell and an inner hemispherical geometry to suit the varying modular head diameters. Inserts/bearings are inserted into the acetabular shell intra-operatively and are available in varying sizes to match the acetabular shell diameters. The insert/bearings are available in Biolox Delta ceramic (CeramTec AG).
  Arms: Hip implant2

SUMMARY:
Evaluate the safety and effectiveness of patients who received G7 Acetabular system in conjunction with Ceramic on Ceramic articulation and Taperloc Complete Microplasty stem compared to patients who received the Exceed ABT Acetabular system with the same combination

DETAILED DESCRIPTION:
This study will be a multi-center randomized controlled study. Eligible patients will be randomly assigned to receive a combination of G7 Acetabular system with CoC articulation and Taperloc Complete Microplasty stem or Exceed ABT Acetabular system with CoC articulation and Taperloc Complete Microplasty stem. Patient demographics, preoperative clinical outcomes, operative information, postoperative clinical outcome, radiographic assessment, incidence of squeaking, incidence of dislocation, implant survivorship and adverse events will be collected prospectively.

ELIGIBILITY:
Inclusion Criteria:

1. Non-inflammatory degenerative joint disease, including osteoarthritis and avascular necrosis.
2. Rheumatoid arthritis.
3. Correction of functional deformity.
4. Treatment of non-union, femoral neck fracture, and trochanteric fractures of the proximal femur with head involvement, unmanageable by other techniques.
5. Revision of previously failed total hip arthroplasty.
6. age over 20 years old

Exclusion Criteria:

1. uncooperative patient or patient with neurologic disorders who are incapable of following directions,
2. osteoporosis,
3. metabolic disorders which may impair bone formation,
4. osteomalacia,
5. distant foci of infections which may spread to the implant site,
6. rapid joint destruction, marked bone loss or bone resorption apparent on roentgenogram, and
7. vascular insufficiency, muscular atrophy, or neuromuscular disease.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2015-05; Primary Completion 2016-06 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
the safety and effectiveness of patients (Harris Hip Score) | 1 year
  Harris Hip Score

SECONDARY OUTCOMES:
Gruen zone analysis | Immediate post-op, 6 months, 1 year, 2 year
  Gruen zone analysis of the femoral component and Charnley-DeLee zone analysis of the acetabular system
Loosening on its implant | Immediate post-op, 6 months, 1 year, 2 year
  The presence of signs of loosening on its implant
Squeaking sounds | 6 months, 1 year, 2 year
  Number of patients with squeaking Sounds
Dislocation | 6 months, 1 year, 2 year
  Dislocation at different follow-up visits

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Joon Yoo, Ph.D, Principal Investigator — Seoul Nat'l Univ. Hospital; Kee-Hyung Rhyu, Ph.D, Principal Investigator — Kyung Hee Uni. Hospital at Gangdong; Seung-Jae Lim, Ph.D, Principal Investigator — Samsung Medical Center; Seung-Bum Han, Ph.D, Principal Investigator — Korea Uni. Anam Hospital
Locations (3):
- South Korea (3):
  - Kyunghee Univ. Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Korea Univ. Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-08): https://cdn.clinicaltrials.gov/large-docs/90/NCT02340390/Prot_SAP_000.pdf